CLINICAL TRIAL: NCT06090084
Title: Investigation of the Musculoskeletal and Respiratory System Factors Affecting Functional Capasity in Multiple Sclerosis
Brief Title: Investigation of Factors Affecting Functional Capasity in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Gözde KAYA, Research Assistant, Izmir Bakircay University
Other Study IDs: 839-819
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis: Multiple sclerosis patients
  Interventions: Other: Evaluation
- Healthy Controls: Healthy subjects
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Functional capacity, balance, core muscle strength, trunk muscle structure, lower extremity muscle strength, upper extremity functions, fatigue and respiratory muscle strength will be evaluated.

SUMMARY:
Functional exercise capacities of Multiple Sclerosis (MS) patients decrease with the effect of symptoms and sedentary lifestyle. A decrease in aerobic capacity may be manifested by a decrease in walking distance or speed, or by restriction in activities of daily living. Decreased aerobic capacity is associated with many factors such as increased risk of cardiovascular disease, decline in cognitive functions, and decreased health-related quality of life. In this respect, measurement of aerobic capacity is one of the important physiological measurements in terms of evaluating the existing functional status of individuals and preparing rehabilitation programs appropriately for individuals. According to studies in the literature, functional capacity in MS patients has been found to be associated with many individual and disease-related factors. However, studies on musculoskeletal and respiratory system factors that may affect functional capacity are insufficient in number. The aim of this study is to examine the effects of balance, core muscle strength, trunk muscle structure, lower extremity muscle strength, upper extremity functions, fatigue and respiratory muscle strength on the functional capacities of MS patients.

Functional capacities of MS patients who met the inclusion criteria will be evaluated with the 6-Minute Walk Test, balance assessments with the Mini Balance Evaluation Systems Test, the strength of the core muscles with the pressurize biofeedback unit, the thickness of the trunk muscles by the Ultrasound Imaging Method, the muscle strength of the lower extremities with the 5 Times Sit to Stand Test, for upper extremity functions, grip strength will be evaluated with a hand dynamometer and Arm Functions Questionnaire in Multiple Sclerosis, fatigue with the Fatigue Severity Scale and respiratory muscle strength will be evaluated by measuring Maximal Inspiratory Pressure and Maximal Expiratory Pressure with an electronic pressure transducer.

The cumulative effects of the parameters to be evaluated on functional capacity in MS patients will be examined by multivariate linear regression analysis and the cumulative total variance will be obtained in terms of R2. Investigation of musculoskeletal system factors that may affect functional capacity and determining which factor contributes more will benefit clinicians and researchers working in this field in terms of evaluating patients and establishing rehabilitation programs.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory disease of unknown etiology, characterized by demyelination, myelin damage, axonal loss and gliosis in the Central Nervous System (CNS). MS symptoms vary depending on the affected area in the CNS. Some of the clinical symptoms are: spasticity, fatigue, loss of muscle strength, tremor, balance problems, exercise intolerance, pain, sensory disorders, bladder and bowel problems, cognitive disorders, depression and sleep disorders. The symptoms seen in MS disease negatively affect the daily life activities of individuals and cause a decrease in their quality of life.

Cardiopulmonary fitness relates to the ability to perform dynamic, moderate to high-intensity exercise of large muscle groups for extended periods of time.

Performance in this type of exercise depends on the functional state of the cardiovascular, respiratory and musculoskeletal systems. Functional exercise capacity in MS patients is impaired compared to healthy individuals and is significantly associated with factors at all levels of the International Classification of Functioning, Disability and Health (ICF) model. A decrease in aerobic capacity may manifest itself as a decrease in walking distance or speed or a limitation in daily living activities. Decreased aerobic capacity is associated with many factors such as increased risk of cardiovascular disease, decline in cognitive functions and decrease in health-related quality of life. In this respect, aerobic capacity measurement is one of the important physiological measurements in terms of evaluating the existing functional status of individuals and preparing rehabilitation programs appropriately for individuals.

According to studies in the literature, functional capacity in MS patients has been found to be related to many individual-specific and disease-related factors. In addition, examining the musculoskeletal system factors that may affect functional capacity and investigating their contributions to functional capacity will be guiding in planning the rehabilitation programs of patients.

Studies investigating factors affecting functional capacity in MS patients are insufficient in number. In our study, the contributions of balance, core muscle strength, trunk muscle structure and upper extremity functions to functional capacity in MS patients will be investigated. Many factors that may be related to functional capacity have been investigated in the literature. However, it has been seen that there is a need for studies on the effects of these factors on functional capacity using regression models.

The aim of this study is to examine the effects of balance, core muscle strength, trunk muscle structure, lower extremity muscle strength, upper extremity functions, fatigue and respiratory muscle strength on the functional capacities of MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years.
* Having MS diagnosed by a neurologist.
* Having a maximum score of 6.5 on the Expanded Disability Status Scale (EDSS).
* No change in medication in the last 6 months.
* Not having had an attack in the last 3 months.
* To be able to walk 100 meters independently
* To be able to read and write

Exclusion Criteria:

* Having another non-MS health problem that would preclude evaluations.
* Having a peripheral vestibular problem.
* Having a cardiopulmonary or orthopedic problem.
* Having a mental problem
* To have received physiotherapy and rehabilitation in the last 3 months.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis patients and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test (6MWT) | The evaluation will take approximately 10 minutes.
  The 6-minute walk test will be performed according to the procedure of Goldman et al. (2008).

SECONDARY OUTCOMES:
The Mini Balance Evaluation Systems Test (Mini BESTest) | The evaluation will take approximately 15 minutes.
  The Mini Balance Evaluation Systems Test (Mini BESTest) will be used in the evaluation of balance. Mini BESTest consists of 4 sub-titles, namely preparatory movement, reactive postural control, sensory orientation and dynamic walking, and a total of 14 items. Each subheading has its own overall rating. The total score of the preparatory movement, reactive postural control and sensory orientation is 6, and the total score of the dynamic walking subheading is 10. The highest score that can be obtained from the test is 28. As the score decreases, the physical condition worsens.
Evaluation of Core Muscles Strength | The evaluation will take approximately 15 minutes.
  Pressure biofeedback device will be used to evaluate the activity of Transversus Abdominis (TrA) and Multifidus (M) muscles.
Evaluation of Trunk Muscle Structure | The evaluation will take approximately 20 minutes.
  Trunk musculature will be examined using ultrasound imaging of the lateral abdominals (transversus abdominis, internal oblique, external oblique) and multifidus muscles.
5 Times Sit To Stand Test | The evaluation will take approximately 3 minutes.
  The 5 times sit to stand test will be used to evaluate the general muscle strength of the lower extremity. It has been shown that this test gives information about the lower extremity muscle strength of MS patients. First, the participants are explained how the test is administered. Then the test is shown once. The participant, who sits in a chair with a height of 45 cm and a depth of 41 cm, without arm support, is told to stand up and sit down 5 times, not to sit back until their knees are fully extended each time they stand up, and to do the test as fast as they can. Before the test begins, participants are asked to place their arms crossed over their chest and maintain this position throughout the test. The test is repeated 3 minutes after the first application. The test result, which is completed in a shorter time than the results of these two applications, is used for statistical analysis. Time recording will be made with a manually controlled electronic stopwatch.
Evaluation of Grip Force | The evaluation will take approximately 5 minutes.
  Jamar® hydraulic hand dynamometer will be used to measure the grip force.
The Arm Function in Multiple Sclerosis Questionnaire (AMSQ) | The evaluation will take approximately 5 minutes.
  The Arm Function in Multiple Sclerosis Questionnaire is an MS-specific scale developed to evaluate upper extremity functions. It evaluates the limitation in activities of daily living related to arm function in the last 2 weeks in MS. The total score is obtained by adding up all the scores. The minimum score that can be obtained from the questionnaire is 31 points, and the maximum score is 186 points. As the score increases, the level of functionality decreases.
Fatigue Severity Scale | The evaluation will take approximately 5 minutes.
  It will be used to evaluate the severity of fatigue. The scale has been shown to be valid and reliable in MS patients and in the Turkish population. It consists of 9 items. The Fatigue Severity Scale score is calculated by adding the scores of answers ranging from 1 to 7 given to nine items and averaging them. A high score indicates that the severity of fatigue increases.
Respiratory Muscle Strength Measurement | The evaluation will take approximately 15 minutes.
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be evaluated using an electronic pressure transducer. Respiratory muscle strength assessment will be done by spirometry according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. Maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) will be measured for assessment of respiratory muscles. The tests will be performed in a sitting position using a nose clip. The best of three successful measurements made will be recorded for further analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yeşim Bakar, Principal Investigator — İzmir Bakırçay University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Langeskov-Christensen M, Heine M, Kwakkel G, Dalgas U. Aerobic capacity in persons with multiple sclerosis: a systematic review and meta-analysis. Sports Med. 2015 Jun;45(6):905-23. doi: 10.1007/s40279-015-0307-x. PMID 25739555
- [Background] Freund JE, Stetts DM, Vallabhajosula S. Relationships between trunk performance, gait and postural control in persons with multiple sclerosis. NeuroRehabilitation. 2016 Jun 30;39(2):305-17. doi: 10.3233/NRE-161362. PMID 27372366
- [Background] Wetzel JL, Fry DK, Pfalzer LA. Six-minute walk test for persons with mild or moderate disability from multiple sclerosis: performance and explanatory factors. Physiother Can. 2011 Spring;63(2):166-80. doi: 10.3138/ptc.2009-62. Epub 2011 Apr 13. PMID 22379256